CLINICAL TRIAL: NCT02842398
Title: Independent Walking Speed and Crossing a City Street
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Blythedale Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Balance_Master
Record Dates: First submitted 2016-07-18; First posted 2016-07-22 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Balance Problems; Cerebral Palsy
Keywords: gait; balance; street-crossing
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Balance Master Training (Experimental): Children receive one weekly Balance Master training session, in addition to their weekly physical therapy sessions. During Balance Master training, children practice balance on a Balance Master device that simulates crossing a city street.
  Interventions: Behavioral: Balance Master
- Customary Care (Active Comparator): Children received their customary scheduled physical therapy sessions, without Balance Master training
  Interventions: Behavioral: Customary Care

INTERVENTIONS:
Behavioral: Balance Master
  Arms: Balance Master Training
Behavioral: Customary Care
  Arms: Customary Care

SUMMARY:
The purpose of this study is to determine if selected sequence training using the Balance Master, added to established physical therapy treatment programs, will increase gait velocity of ambulatory children receiving inpatient or outpatient rehabilitation in relation to their ability to cross an intersection within the confines of community traffic signal (>120 cm/sec).

DETAILED DESCRIPTION:
The ability to adequately perform functional tasks at a level that allows independent community living is key to measuring the success of any physical therapy program. The essential tasks needed to allow independent community living have been well documented in the elderly population. However, these tasks have not been delineated in the pediatric population. The investigators aim to determine if selected sequence training using the Balance Master, added to established physical therapy treatment programs, will increase gait velocity of ambulatory children receiving in-or outpatient rehabilitation in relation to their ability to cross an intersection within the confines of community traffic signal (>120 cm/sec). One essential task that is necessary in the urban environment is to have the ability to cross a street within the time constraint of a traffic signal. Walking speed becomes increasingly important for those living in urban settings, as the ability to cross the street safely is fundamental for achieving independence. One of the major criticisms of clinic/lab-based measures of gait speed is that relative performance may not be representative of independence within the community. Participants aged 5 to 21 years, will be recruited from the patient population at Blythedale Children's Hospital for a six week trial. Children will be assigned to one of two random groups: one weekly Balance Master sequence training group (in addition to their regularly scheduled therapy sessions) and a group that continue regularly scheduled therapy sessions alone. Gait velocity will be measured by "Walk Across" Functional Assessment using Balance Master long force plate.

ELIGIBILITY:
Inclusion Criteria:

* Ability to ambulate independently at least 25 feet with or without assistance device and/or orthoses.
* Receiving physical therapy services that include ambulation training.

Exclusion Criteria:

* Diagnosis of a progressive disorder.
* Inability to follow directions.
* Uncorrected vision impairment.
* Require additional physical assistance to ascend a ramp and over force plate.
* Refusal to participate.

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2010-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in gait velocity after intervention | measured at day 1 of intervention and end of week 6 of intervention
  Measure gait velocity as participant walks across a force plate on the floor

SECONDARY OUTCOMES:
Weight | Day 1 of Intervention
  Body weight on a digital scale

CONTACTS AND LOCATIONS:
Locations (1):
- Blythedale Children's Hospital, Valhalla, New York, United States